CLINICAL TRIAL: NCT03299400
Title: Continuous Intraocular Pressure Patterns in Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kenny Kwan, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UW 16-207
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Intraocular Pressure
Keywords: IOP

STUDY DESIGN:
Intervention Model Description: All eligible patients who have given informed consent will attend the ophthalmology clinic for screening.
  Patient will undergo general anaesthesia for prone spinal surgery. The degree of inclination was set prior to the start of the case and independently confirmed using a goniometer. Patients will be placed in the prone position on a Jackson Spine table.
  Once positioned, the head is carefully placed on the GentleTouch prone positioning pillow of the appropriate size.
  Patient will continue to wear the contact lens postoperatively for a total of 24 hours or until the patient cannot tolerate the contact lens. After removal of the contact lens sensor, the recorded profiles will be collected and visualized graphically on a computer interface. The output of the sensor expressed in voltage, and can be analysed in real time points corresponding to the intraoperative events.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Contact lens sensor (Experimental): Patient will continue to wear the contact lens postoperatively for a total of 24 hours or until the patient cannot tolerate the contact lens. After removal of the contact lens sensor, the recorded profiles will be collected and visualized graphically on a computer interface.
  Interventions: Device: Contact lens sensor

INTERVENTIONS:
Device: Contact lens sensor — Patient will continue to wear the contact lens postoperatively for a total of 24 hours or until the patient cannot tolerate the contact lens. After removal of the contact lens sensor, the recorded profiles will be collected and visualized graphically on a computer interface.

SUMMARY:
Post-operative visual loss is a rare but serious complication after surgery. It is most significantly correlated with prone spinal surgery with a prolonged duration. The cause and risk factors are not elucidated, but the majority of the cases are due posterior ischaemic optic neuropathy (PION). This entity is directly related to the ocular perfusion pressure (OPP), which is estimated as the difference between mean arterial blood pressure (MAP) and intraocular pressure (IOP). Autoregulation is believed to maintain a constant perfusion to the optic nerve despite fluctuations in the perfusion pressure.

IOP is known to increase in the prone position thus putting susceptible patients at risk for inadequate ocular nerve perfusion. Most of the evidence comes from animal and healthy volunteer studies and cannot give an accurate insight into the subtle changes of intra-operative IOP. All the published studies employed the use of a tonometer, which may have rooms for measurement errors due to inadvertent pressure on the globe while retracting the eyelids, particularly when there is significant periorbital/conjunctival swelling in the prone position. The majority of the studies recruited healthy volunteers in a simulated surgical setting so other fluctuating parameters, which can affect intraoperative IOP, cannot be measured. In the few reports where patients undergoing surgery in the prone position were studies, IOP measurements were taken at non-continuous monitoring at time intervals, thus the effects of changes in blood volume, MAP, central venous pressure (CVP) and PaCO 2 could not be studied. Lastly, all the literature consists of case series only with no control group so the effect of position cannot be evaluated independently of the other factors.

The investigators therefore propose to conduct a prospective study with continuous intraoperative IOP monitoring to give us further insight into the physiological changes of IOP in patients undergoing spine surgery, and identify the risk factors related to fluctuations of IOP during prone spinal surgery.

DETAILED DESCRIPTION:
Post-operative visual loss (POVL) is a rare but serious complication after surgery.

One of the known associations is prone spinal surgery with a prolonged duration.

The cause is not completely understood, but some of the risk factors for developing POVL include anaemia, hypotension, the duration of surgery and patient factors such as age, hypertension and atherosclerosis. There are also some unidentifiablerisk factors that may predispose young healthy patients to POVL. Once the patient develops POVL, it is usually irreversible, and the patient is left with a permanent disability.

The majority of POVL cases that occur with prone spinal surgery are due to posterior ischaemic optic neuropathy (PION). PION is directly related to the ocular perfusion pressure (OPP), which is estimated as the difference between mean arterial blood pressure (MAP) and intraocular pressure (IOP). Autoregulation is believed to maintain a constant perfusion to the optic nerve despite fluctuations in the perfusion pressure.

However, there is a knowledge gap in the physiological changes of IOP during prone surgery. IOP is a highly dynamic parameter, and the most widely used method to measure it is using a handheld tonometer. The main limitation of this technique is the isolated nature of its measurements, as it can only be taken at regular intervals, and may not reflect the full range of IOP changes. Studies on IOP during prone position in the current literature have all used this technique. 1-5 Hence subtle changes of IOP can be undetected, as interval measurements cannot reflect short-term variations that occur within seconds or minutes. Furthermore, most of the studies are performed on animals or healthy volunteers 5,6 , which further limit the interpretation of their results. For the few studies performed on anaesthetised patients undergoing spinal surgeries, the duration of surgery is short or mixed, so the critical time point may not have been studied. The American Society of Anesthesiologists Postoperative Visual Loss Registry suggests that an anaesthetic duration of greater than 6 hours is more correlated with POVL.

Using state of the art technology Over the past five years, advances in technology have led to the development of devices that allow 24 hour continuous IOP monitoring. The new system makes use of microelectromechanical systems, nanotechnology, and telemetry to allow continuous monitoring. A disposable contact lens sensor, first proposed by Leonardi et al. 8 , is now commercially available (SENSIMED Triggerfish; Sensimed AG, Lausanne, Switzerland). This technology can acquire data points over a 24 hour period corresponding to 30 seconds of continuous measurements. It measures changes in the ocular dimensions at the corneoscleral junction, which corresponds to changes to IOP and volume. The microprocessor within the lens transmits data to an external antenna, and the profiles can be stored in a portable recorder. 9 Although this sensor does not measure IOP directly, it gives measurements with a composite of IOP and volume changes, and it is most valuable in documenting relative changes of IOP-related events and their timing. It is also well tolerated in real life patients, and have been used to document IOP changes in patients with glaucoma and thyroid eye disease. 9-11 This is the only non-invasive temporary continuous monitoring in the system that can be used in human beings. This new technology is therefore ideal in detecting subtle changes in IOP pattern in prone spinal surgery. It will provide a continuous monitoring which can be correlated with the patient's level of anaesthesia, arterial pressure fluctuations and volume status, and can contribute to improved understanding of IOP changes during prone spinal surgery, which may in turn bridge the knowledge gap of the causes of POVL.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age 18 to 80 years inclusive
* No pre-existing eye pathology (excluding refractive error), patients with glaucoma, history of eye injury or ophthalmic surgery
* No known allergy to contact lens material
* Patients undergoing anterior cervical spine surgery and prone spine surgery for duration of 3 hours or longer

Exclusion Criteria:

* Unable to comply with follow up or give informed consent
* Cannot tolerate wearing contact lens
* Has active eye infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Report the physiological changes of IOP patterns during prone spinal surgery | 1 year
  The outcome measure will be to report the physiological changes of IOP patterns during prone spinal surgery.

SECONDARY OUTCOMES:
Correlate any intraoperative risk factors that may cause IOP fluctuations | 1 year
  To correlate any intraoperative risk factors that may cause IOP fluctuations
Documentation of IOP changes after the surgery until the contact lens sensor is removed | 1 year
  Documentation of IOP changes after the surgery until the contact lens sensor is removed

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kenny Kwan, BMBCh(Oxon), Principal Investigator — The University of Hong Kong
Locations (1):
- Duchess of Kent Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carey TW, Shaw KA, Weber ML, DeVine JG. Effect of the degree of reverse Trendelenburg position on intraocular pressure during prone spine surgery: a randomized controlled trial. Spine J. 2014 Sep 1;14(9):2118-26. doi: 10.1016/j.spinee.2013.12.025. Epub 2014 Jan 20. PMID 24456677
- [Background] Sugata A, Hayashi H, Kawaguchi M, Hasuwa K, Nomura Y, Furuya H. Changes in intraocular pressure during prone spine surgery under propofol and sevoflurane anesthesia. J Neurosurg Anesthesiol. 2012 Apr;24(2):152-6. doi: 10.1097/ANA.0b013e31823fe822. PMID 22274735
- [Background] Yoshimura K, Hayashi H, Tanaka Y, Nomura Y, Kawaguchi M. Evaluation of predictive factors associated with increased intraocular pressure during prone position spine surgery. J Anesth. 2015 Apr;29(2):170-4. doi: 10.1007/s00540-014-1921-8. Epub 2014 Sep 24. PMID 25249431
- [Background] Deniz MN, Erakgun A, Sertoz N, Yilmaz SG, Ates H, Erhan E. The effect of head rotation on intraocular pressure in prone position: a randomized trial. Braz J Anesthesiol. 2013 Mar-Apr;63(2):209-12. doi: 10.1016/j.bjane.2012.03.008. Epub 2013 Aug 13. PMID 24565128
- [Background] Walick KS, Kragh JE Jr, Ward JA, Crawford JJ. Changes in intraocular pressure due to surgical positioning: studying potential risk for postoperative vision loss. Spine (Phila Pa 1976). 2007 Nov 1;32(23):2591-5. doi: 10.1097/BRS.0b013e318158cc23. PMID 17978659
- [Background] Setogawa A, Kawai. Measurement of intraocular pressure by both invasive and noninvasive techniques in rabbits exposed to head-down tilt. Jpn J Physiol. 1998 Feb;48(1):25-31. doi: 10.2170/jjphysiol.48.25. PMID 9538286
- [Background] Postoperative Visual Loss Study Group. Risk factors associated with ischemic optic neuropathy after spinal fusion surgery. Anesthesiology. 2012 Jan;116(1):15-24. doi: 10.1097/ALN.0b013e31823d012a. PMID 22185873
- [Background] Leonardi M, Pitchon EM, Bertsch A, Renaud P, Mermoud A. Wireless contact lens sensor for intraocular pressure monitoring: assessment on enucleated pig eyes. Acta Ophthalmol. 2009 Jun;87(4):433-7. doi: 10.1111/j.1755-3768.2008.01404.x. Epub 2008 Nov 12. PMID 19016660
- [Background] Mansouri K, Weinreb R. Continuous 24-hour intraocular pressure monitoring for glaucoma--time for a paradigm change. Swiss Med Wkly. 2012 Mar 28;142:w13545. doi: 10.4414/smw.2012.13545. eCollection 2012. PMID 22457163
- [Background] Parekh AS, Mansouri K, Weinreb RN, Tafreshi A, Korn BS, Kikkawa DO. Twenty-four-hour intraocular pressure patterns in patients with thyroid eye disease. Clin Exp Ophthalmol. 2015 Mar;43(2):108-14. doi: 10.1111/ceo.12400. Epub 2014 Sep 29. PMID 25132194
- [Background] De Smedt S, Mermoud A, Schnyder C. 24-hour intraocular pressure fluctuation monitoring using an ocular telemetry Sensor: tolerability and functionality in healthy subjects. J Glaucoma. 2012 Oct-Nov;21(8):539-44. doi: 10.1097/IJG.0b013e31821dac43. PMID 21602707